CLINICAL TRIAL: NCT02227732
Title: A Pilot Study Evaluating the Safety and Effectiveness of a New Pleural Catheter for the Medical Management of Symptomatic, Recurrent, Malignant Pleural Effusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-IS-VH-13-001; CI20130054 (Other: UK MHRA)
Record Dates: First submitted 2014-07-08; First posted 2014-08-28 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Malignant Pleural Effusions
MeSH Terms: conditions — Pleural Effusion, Malignant

ARMS (1):
- New Indwelling Pleural Catheter (Other)
  Interventions: Device: New Indwelling Pleural Catheter

INTERVENTIONS:
Device: New Indwelling Pleural Catheter — Placement of an indwelling catheter in the pleural space. Drainage of effusions until resolution.

SUMMARY:
The purpose of this study is to determine whether a new catheter is safe and effective in treating malignant pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject has a symptomatic malignant pleural effusion requiring intervention. For an effusion to be defined as malignant, at least one of the following must be true:

   * There is histocytological confirmation of pleural malignancy
   * The effusion is an exudate (as per Light's criteria) in the context of histocytologically proven malignancy elsewhere, with no other clear cause for fluid identified
3. Subject has a history of at least one ipsilateral pleural effusion causing dyspnoea that responded to thoracentesis where the lung expanded and the dyspnoea was relieved.
4. Subject is willing and able to provide written informed consent.
5. Subject is willing and able to meet all study requirements, including attending follow-up visits or receiving trial-related telephone calls.
6. There is sufficient fluid on thoracic ultrasound to allow safe insertion of an indwelling pleural catheter
7. Negative pregnancy test if appropriate

Exclusion Criteria:

1. Subject has significant trapped lung (>20%), or a proximal bronchial obstruction which is likely to lead to trapped lung.
2. Subject has a Karnofsky score of less than 50, or a WHO/ECOG performance status of 3* or more.
3. Subject is pregnant, planning to become pregnant, or is lactating.
4. Subject has a history of empyema.
5. Subject has a history of chylothorax.
6. Subject has an uncorrected coagulopathy.
7. Subject is allergic to device materials.
8. Subject has evidence, in the opinion of the Chief Investigator, of either on-going systemic or pleural infection.
9. Subject has had a lobectomy or pneumonectomy on the side of the effusion.
10. Subject has undergone a previous attempt at pleurodesis which has failed.
11. Subject has previously been diagnosed with a serious immunodeficiency disorder.
12. Subject has bilateral pleural effusions, with both being at least moderate in size (greater than 1/3 of the hemithorax on chest x-ray).
13. Subject has evidence of fluid loculation such that attempts at pleurodesis are likely to be futile.
14. Subject has a mediastinal shift of ≥2cm toward the side of the effusion.
15. Subject is receiving concurrent intrapleural chemotherapy or radiation therapy to the ipsilateral chest.
16. Subject has any clinical condition, diagnosis, or social circumstance that, in the opinion of the Chief Investigator, would mean participation in the study would be contraindicated.
17. Subject has no access to a telephone
18. No details of blood values (full blood count, clotting screen, urea and electrolytes, liver function) from within the last 10 days * Patients who have a performance status of 3 may be considered for the trial if the removal of their fluid would likely improve their performance score by 1 or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Device -related safety and the number of adverse events. | 28 days post catheter insertion

SECONDARY OUTCOMES:
pleurodesis success | 14 days
  Assessed by chest x-ray, thorachic ultrasound, and confirmation the catheter is patent.
Pleurodesis success | 28 days
  Assessed by chest x-ray, thoracic ultrasound and confirmaiton the catheter is patent.
pleurodesis success | 60 days
  Assessed by chest x-ray, thoracic ultrasound and confirmaiton the catheter is patent.

OTHER OUTCOMES:
Breathlesness | 14, 28, 60 days
Chest Pain | 14, 28, 60 days
Time to pleurodesis | 14, 28, 60 days
Quality of Life | 14, 28, 60 days
Need for further pleural intervention post catheter removal | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Southmead Hospital - Academic Resporatory Unit, Westbury on Severn, Bristol, United Kingdom